CLINICAL TRIAL: NCT03932474
Title: DOUBLE BLIND, RANDOMIZED, PLACEBO CONTROLLED STUDY TO EVALUATE THE EFFICACY OF SAMEUP IN SUBJECTS CHARACTERIZED BY MILD TO MODERATE DEPRESSION SYMPTOMS
Brief Title: EVALUATION OF EFFICACY OF SAMEUP IN SUBJECTS WITH DEPRESSION SYMPTOMS: A RANDOMIZED STUDY
Acronym: SAMEUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutrilinea srl (Industry)
Collaborators: Hippocrates Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAMEUP
Record Dates: First submitted 2019-04-19; First posted 2019-04-30 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Depressive Symptoms
Keywords: depression; probiotic; SAMe; Lactobacillus plantarum 299v; anxiety; insomnia; irritable bowel syndrome; randomized controlled study
MeSH Terms: conditions — Depression; Anxiety Disorders; Sleep Initiation and Maintenance Disorders; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAMEUp (Experimental): SAMEUp, the Investigational Food Supplement (IFS), is an oral formulation (tablet) containing S-adenosyl methionine (SAMe) 200 mg and Lactobacillus plantarum HEAL9 1x109 CFU.
  Interventions: Combination Product: SAMEUp
- Placebo (Placebo Comparator): Placebo is an oral formulation of inert tablet. Placebo and SAMEUp are identical in shape, size, colour and taste.
  Interventions: Other: Placebo

INTERVENTIONS:
Combination Product: SAMEUp — One tablet per day of food supplements containing S-adenosyl methionine (SAMe) 200 mg and Lactobacillus plantarum HEAL9 1x109 CFU.
  Arms: SAMEUp
Other: Placebo — One tablet per day identical in shape, size, colour and taste to the SAMEUp tablet
  Arms: Placebo

SUMMARY:
This study is planned to assess the efficacy of SAMEUp versus placebo after six weeks of treatment in subjects characterized by depression symptoms according to ICD-10 (International Classification of Diseases - 10th revision) diagnostic criteria and confirmed by mean of Zung's Self-Rating Depression Scale.

DETAILED DESCRIPTION:
Depression is a common condition of low mood and aversion to activity that can affect a person's thoughts, behaviour, tendencies, feelings, and sense of well-being.

Several literature findings suggest that an oral combination of the two food supplements SAMe (S-adenosyl-L-methionine) and probiotic Lactobacillus plantarum might be favourable in relieving some of symptoms of depression, particularly in the mild to moderate forms of this condition. This double blind placebo controlled clinical study aims to evaluate this hypothesis. In particular, the primary objective is to assess, versus placebo, the efficacy of SAMEUp in improving the overall symptomology of depression after 6 weeks of treatment. Subjects with mild to moderate depression were identified according to ICD-10 diagnostic criteria and confirmed by mean of Zung's Self-Rating Depression Scale.

SAMEUp, the investigational food supplement, is an oral formulation (tablet) containing S-adenosyl methionine (SAMe) 200 mg and Lactobacillus plantarum HEAL9 1x109 CFU, already notified to the Ministry of Health as food supplement.

Placebo is an oral formulation of inert tablet. Placebo and SAMEUp are indistinguishable.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent, personally signed and dated by the subject.
2. Males and females, aging 18-60 years old (limits included).
3. Diagnosis of mild to moderate recurrent depressive disorder according to the ICD-10 / F33 criteria (World Health Organization, 2004).
4. Subject who, having completed the Z-SDS depression questionnaire, has a raw score between 41 and 55 (including limits).
5. Subject able to comprehend the full nature and purpose of the study, available to cooperate with the Investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Pregnant or breast-feeding woman.
2. Subject with one or more psychiatric disturbances, such as: alcoholism, substance abuse or dependency disorder, bipolar disorder, schizophrenia, or other personality disorder.
3. Subject with known or potential hypersensitivity to any ingredient in the study product.
4. Subject in treatment with psycholeptic drug, such as: antipsychotics, anxiolytics, hypnotics and sedatives.
5. Subject who has taken during the 2 weeks prior to inclusion, who is currently taking or plans to take other orally administered food supplements except the study product. Only multivitamins, salts and trace elements are accepted

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2018-11-20 (Actual)

PRIMARY OUTCOMES:
Improvement in the overall depression symptomatology assessed by the Zung's Self-Rating Depression Scale | 6 weeks
  Absolute change from baseline to six treatment-week of the total score of the Zung's Self-Rating Depression Scale

SECONDARY OUTCOMES:
Improvement in the overall depression symptomatology assessed by the Zung's Self-Rating Depression Scale | 2 weeks
  Absolute change from baseline to two treatment-week of the total score of the Zung's Self-Rating Depression Scale
Improvement in the core depression symptomatology assessed by Zung's Self-Rating Depression Scale | 2 weeks
  Absolute change from baseline to two treatment-week of the core depressive factor of the Zung's Self-Rating Depression Scale.
Improvement in the core depression symptomatology assessed by Zung's Self-Rating Depression Scale | 6 weeks
  Absolute change from baseline to six treatment-week of the core depressive factor of the Zung's Self-Rating Depression Scale.
Improvement in the patient's cognition assessed by Zung's Self-Rating Depression Scale | 2 weeks
  Absolute change from baseline to two treatment-week of the cognitive factor of the Zung's Self-Rating Depression Scale.
Improvement in the patient's cognition assessed by Zung's Self-Rating Depression Scale | 6 weeks
  Absolute change from baseline to six treatment-week of the cognitive factor of the Zung's Self-Rating Depression Scale.
Improvement in the anxiety condition assessed by Zung's Self-Rating Depression Scale | 2 weeks
  Absolute change from baseline to two treatment-week of the anxiety factor of the Zung's Self-Rating Depression Scale.
Improvement in the anxiety condition assessed by Zung's Self-Rating Depression Scale | 6 weeks
  Absolute change from baseline to six treatment-week of the anxiety factor of the Zung's Self-Rating Depression Scale.
Improvement in the somatic condition assessed by Zung's Self-Rating Depression Scale | 2 weeks
  Absolute change from baseline to two treatment-week of the somatic factor of the Zung's Self-Rating Depression Scale.
Improvement in the somatic condition assessed by Zung's Self-Rating Depression Scale | 6 weeks
  Absolute change from baseline to six treatment-week of the somatic factor of the Zung's Self-Rating Depression Scale.
Improvement in the overall symptomatology of depression assessed by Zung's Self-Rating Depression Scale | 2 weeks
  Absolute change from baseline to two treatment-week of the total score of the Zung's Self-Rating Anxiety Scale.
Improvement in the overall symptomatology of depression assessed by Zung's Self-Rating Depression Scale | 6 weeks
  Absolute change from baseline to six treatment-week of the total score of the Zung's Self-Rating Anxiety Scale.
Improvement in the insomnia condition evaluated through the Insomnia Severity Index | 2 weeks
  Absolute change from baseline to two treatment-week of the total score of the Insomnia Severity Index.
Improvement in the insomnia condition evaluated through the Insomnia Severity Index | 6 weeks
  Absolute change from baseline to six treatment-week of the total score of the Insomnia Severity Index.
Improvement in IBS (Irritable Bowel Syndrome) symptoms evaluated through the IBS questionnaire | 2 weeks
  Absolute change from baseline to two treatment-week of the total score of the IBS questionnaire.
Improvement in IBS symptoms evaluated through the IBS questionnaire | 6 weeks
  Absolute change from baseline to six treatment-week of the total score of the IBS questionnaire.
Improvement in the overall health status as measured by the EQ-5D-3L questionnaire | 2 weeks
  Absolute change from baseline to two treatment-week of the EQ-5D-3L questionnaire.
Improvement in the overall health status as measured by the EQ-5D-3L questionnaire | 6 weeks
  Absolute change from baseline to six treatment-week of the EQ-5D-3L questionnaire.
Evaluation of the patient's satisfaction grade | 6 weeks
  Subject's satisfaction grade at the end of the treatment.
Incidence of adverse events described as per frequency and relationship with the study product | 6 weeks
  Adverse events occurrence during the study

CONTACTS AND LOCATIONS:
Locations (1):
- Hippocrates Research, Genoa, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saccarello A, Montarsolo P, Massardo I, Picciotto R, Pedemonte A, Castagnaro R, Brasesco PC, Guida V, Picco P, Fioravanti P, Montisci R, Schiavetti I, Vanelli A. Oral Administration of S-Adenosylmethionine (SAMe) and Lactobacillus Plantarum HEAL9 Improves the Mild-To-Moderate Symptoms of Depression: A Randomized, Double-Blind, Placebo-Controlled Study. Prim Care Companion CNS Disord. 2020 Jun 25;22(4):19m02578. doi: 10.4088/PCC.19m02578. PMID 32589828